CLINICAL TRIAL: NCT02429323
Title: Endotracheal Intubation With Sevoflurane in Surgical Pediatric Patients: Incremental Versus High Concentration Inhalation Induction
Brief Title: Endotracheal Intubation With Sevoflurane in Surgical Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Amir M. Boujan, Senior Anesthesiologist, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 8
Record Dates: First submitted 2015-04-18; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Anesthesia; Reaction
Keywords: induction; pediatrics; sevoflurane; intubation time
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane concentration 8% (Active Comparator): sevoflurane concentration 8% from the start
  Interventions: Drug: Sevoflurane
- incremental sevoflurane (1-8%) (Active Comparator): incremental increase of the concentration each few breaths from 1% to 8%
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — use of 8% sevoflurane in compared to incremental dose increased each few breaths from 1% to 8%
  Other Names: sevorane abbott

SUMMARY:
Aim of the study is to compare the optimal time needed for successful tracheal intubation with immediate 8% sevoflurane and incremental sevoflurane induction in surgical pediatric patients undergoing adenotonsillectomy without using muscle relaxants or opioids

DETAILED DESCRIPTION:
Investigators studied 100 pediatric surgical patients admitted to Sulaimani Teaching Hospital in the Otorhinolaryngology, Head and Neck Surgical Department, from the first of June 2011 to the first of September 2011, Children aged 2-7 years,both genders, ASA physical statuses І and II (ASA I: a healthy normal patient, while ASA II: a patient with mild systemic disease with no functional limitations) were scheduled for elective adenotonsillectomy operations. They were randomly divided into two equal groups according to the induction method.

Group 1 (G1) using incremental induction with sevoflurane (1-8 %) in 100% O2, the vapor concentration is increased by 1% every few breaths.

Group 2 (G2) high concentration of sevoflurane (8%) in 100% O2 from the beginning of induction.

None of them is given premedication or any other adjunct drugs until successful intubation is done; ventilation was assisted and then controlled when possible. If upper airway obstruction occurred, an oropharyngeal airway was immediately inserted. Attempts were made to obtain venous access before laryngoscopy. All patients monitored with electrocardiography (ECG), noninvasive blood pressure monitoring (NIBP), pulse oximetry, and temperature measurements.

Children with extreme weight, suspicion of difficult airway, moved during laryngoscopy, or more than one trial of laryngoscopy needed were excluded from this study.

The endotracheal tube (ETT) size was selected by using the formula (age/4) + 4.5. Only a single laryngoscopy attempt was allowed. Small, brief movements of extremities occurring after (ETT) placement did not considered as exclusion criteria. Anesthesia was delivered by anesthetic machine (Datex Ohmeda), using an Ayer's T-piece with Jackson Ree's modification system, with a fresh gas flow of 6 L/min through a Sevoflurane vaporizer.

Patients were observed until eyelash reflex disappears, pupils centered and constricted. Jaw relaxation and movements were monitored. Ventilation was controlled till the time of laryngoscopy; the vocal cords were completely visible, orotracheal intubation done with Macintosh laryngoscope blade size 2 by the same anesthetist for all the patients. The time from induction until successful tracheal intubation is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-7 years old American society of anesthesiologists physical status class 1 and 2 scheduled for elective adenotonsillectomy operations

Exclusion Criteria:

* Children with extreme weight, suspicion of difficult airway, moved during laryngoscopy, or more than one trial of laryngoscopy needed

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
induction to intubation time in seconds | during the surgery
  effect of high concentration of sevoflurane on shortening the induction to intubation time

CONTACTS AND LOCATIONS:
Overall Officials: Amir M. Boujan, board, Study Director — School of Medicine

REFERENCES:
- [Background] James Duke, Pediatric Anesthesia, Anesthesia Secrets, Philadelphia 2011, Fourth Edition, Chapter 57, Page 396.
- [Background] Johr M. Anaesthesia for tonsillectomy. Curr Opin Anaesthesiol. 2006 Jun;19(3):260-1. doi: 10.1097/01.aco.0000192789.78139.54. No abstract available. PMID 16735808
- [Background] Chawathe M, Zatman T, Hall JE, Gildersleve C, Jones RM, Wilkes AR, Aguilera IM, Armstrong TS. Sevoflurane (12% and 8%) inhalational induction in children. Paediatr Anaesth. 2005 Jun;15(6):470-5. doi: 10.1111/j.1460-9592.2005.01478.x. PMID 15910347
- [Background] Inomata S, Yamashita S, Toyooka H, Yaguchi Y, Taguchi M, Sato S. Anaesthetic induction time for tracheal intubation using sevoflurane or halothane in children. Anaesthesia. 1998 May;53(5):440-5. doi: 10.1046/j.1365-2044.1998.00338.x. PMID 9659016
- [Background] Politis GD, Tobin JR, Morell RC, James RL, Cantwell MF. Tracheal intubation of healthy pediatric patients without muscle relaxant: a survey of technique utilization and perceptions of safety. Anesth Analg. 1999 Apr;88(4):737-41. doi: 10.1097/00000539-199904000-00009. PMID 10195514
- [Background] Redhu S, Jalwal GK, Saxena M, Shrivastava OP. A Comparative Study of Induction, Maintenance and Recovery Characteristics of Sevoflurane and Halothane Anaesthesia in Pediatric Patients (6 months to 6 years). J Anaesthesiol Clin Pharmacol. 2010 Oct;26(4):484-7. PMID 21547175
- [Background] Blair JM, Hill DA, Bali IM, Fee JP. Tracheal intubating conditions after induction with sevoflurane 8% in children. A comparison with two intravenous techniques. Anaesthesia. 2000 Aug;55(8):774-8. doi: 10.1046/j.1365-2044.2000.01470.x. PMID 10947692
- [Background] Fenlon S, Pearce A. Sevoflurane induction and difficult airway management. Anaesthesia. 1997 Mar;52(3):285-6. No abstract available. PMID 9124682
- [Background] Epstein RH, Stein AL, Marr AT, Lessin JB. High concentration versus incremental induction of anesthesia with sevoflurane in children: a comparison of induction times, vital signs, and complications. J Clin Anesth. 1998 Feb;10(1):41-5. doi: 10.1016/s0952-8180(97)00218-3. PMID 9526937
- [Background] Baum VC, Yemen TA, Baum LD. Immediate 8% sevoflurane induction in children: a comparison with incremental sevoflurane and incremental halothane. Anesth Analg. 1997 Aug;85(2):313-6. doi: 10.1097/00000539-199708000-00013. PMID 9249106
- [Background] Dubois MC, Piat V, Constant I, Lamblin O, Murat I. Comparison of three techniques for induction of anaesthesia with sevoflurane in children. Paediatr Anaesth. 1999;9(1):19-23. PMID 10712710